CLINICAL TRIAL: NCT06843291
Title: UNIVERSAL GENETIC TESTING OF PATIENTS WITH HEMATOLOGICAL MALIGNANCIES (UGT)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2218223
Record Dates: First submitted 2025-02-20; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Hematologic Disease
Keywords: Genetic testing; hematological malignancies
MeSH Terms: conditions — Hematologic Diseases; Hematologic Neoplasms | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- genetic testing for hematological malignancies (Experimental): Single arm study for patients with hematological malignancies who agree to genetic testing.
  Interventions: Genetic: Genetic Testing for hematological malignancies

INTERVENTIONS:
Genetic: Genetic Testing for hematological malignancies — combined skin punch biopsy/BM aspiration technique, followed by NGS and OGM.

SUMMARY:
We propose to perform NGS and OGM with DNA extracted from bone marrow (BM; site of cancer) and NGS on skin fibroblast DNA (proxy for germline) on all patients with hematologic malignancies (HM) who undergo a standard-of-care BM biopsy at Georgia Cancer Center/Wellstar MCG Health. Simultaneous 4 mm punch skin biopsy for fibroblast culture will be obtained at the planned puncture site of the BM biopsy. The bone marrow biopsy and aspirate are already part of the patient's scheduled medical evaluation and the punch biopsy of the skin is the only additional procedure involved in the study.

DETAILED DESCRIPTION:
Genetic data is transforming the understanding and management of cancers of all types.

The detection of pathogenic germline genetic variants (mutations) underlying the formation of cancer is important because the genetic information can inform optimal treatment for individuals with cancer and can be used to modify cancer risk in family members who are carriers for the variant but who have not developed cancer. Germline next generation sequencing (NGS) has only recently begun to be used to assess for hereditary risk in hematological malignancies (HM), and in particular beyond myeloid HMs. NGS detects small genetics changes such single base substitutions and small deletions, whereas a new technique called optical genome mapping (OGM) is able to detect large structural genetic changes in tumor DNA. OGM is well established here in Molecular Pathology but has only recently been applied to the study of HMs.

We propose to perform NGS and OGM with DNA extracted from bone marrow (BM; site of cancer) and NGS on skin fibroblast DNA (proxy for germline) on all patients with hematologic malignancies (HM) who undergo a standard-of-care BM biopsy at Georgia Cancer Center/Wellstar MCG Health. Simultaneous 4 mm punch skin biopsy for fibroblast culture will be obtained at the planned puncture site of the BM biopsy. The bone marrow biopsy and aspirate are already part of the patient's scheduled medical evaluation and the punch biopsy of the skin is the only additional procedure involved in the study. We will compare BM and germline variants in order to determine their rate and concordance, examine the percent of germline variants that are likely to be the cause of the HM, assess the impact of the germline finding on treatment choices, and determine the impact of germline findings on family members. New data from OGM will be compared to NGS

ELIGIBILITY:
Inclusion Criteria:

- a. Age ≥ 18 years of age. b. A new diagnosis of HM. c. Diagnostic bone marrow to be performed at Wellstar MCG Health/Georgia Cancer Center.

d. Ability and willingness to provide informed consent in English to undergo skin biopsy for fibroblast culture and NGS for comparison with the BM NGS.

Exclusion Criteria:

* There are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of all patients with hematological malignancies who agree to undergo genetic testing | 5 years
  The primary endpoint will be the percentage of all patients with newly diagnosed HMs who undergo BM/fibroblast DNA NGS testing.

CONTACTS AND LOCATIONS:
Overall Officials: John Henson, MD, Principal Investigator — Medical College of Georgia at Augusta University